CLINICAL TRIAL: NCT04429854
Title: A Randomized, Open-label, Adaptive, Proof-of-concept Clinical Trial of Donated Antibodies Working Against With COVID-19: DAWN-PLASMA
Brief Title: Donated Antibodies Working Against nCoV
Acronym: DAWN-Plasma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Federal Knowledge Centre (KCE) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S63992
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: 483 patients with 2:1 randomization. 320 patients receiving Convalescent Plasma - 163 patients receiving Standard of Care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convalescent Plasma (Experimental): 4 units of convalescent plasma:
  * 2 units of plasma are administered within 12h after randomization, but preferably as soon as practically possible
  * 2 units of plasma should be administered between 24h and 36h after the first infusion
  Interventions: Biological: Convalescent Plasma; Drug: Standard of care
- Standard of Care (Other): Since there are no current approved treatment options for COVID-19, the standard of care is mostly supportive. Since there are no current approved treatment options for COVID-19, the standard of care is mostly supportive.
  Interventions: Drug: Standard of care

INTERVENTIONS:
Biological: Convalescent Plasma — 4 units of convalescent plasma:
  * 2 units of plasma are administered within 12h after randomization, but preferably as soon as practically possible
  * 2 units of plasma should be administered between 24h and 36h after the first infusion
  Other investigational products may be added as part of the adaptive study design.
  Arms: Convalescent Plasma
Drug: Standard of care — Since there are no current approved treatment options for COVID-19, the standard of care is mostly supportive.

SUMMARY:
This a phase II, proof-of-concept study. In the present study, we investigate if the administration of blood-plasma from patients recovered from COVID-19, could be effective to treat patients who are severely ill because of a COVID-19 infection. The general idea behind the transfusion, is that plasma of recovered patients contains antibodies that could eliminate the novel coronavirus causing COVID-19, and lead to a less severe course of the disease, or a faster healing. Simply put, in this study we would like to investigate whether 'borrowed immunity' from a person who has cured from this disease, could be applied to cure other patients more rapidly.

DETAILED DESCRIPTION:
In December 2019, a new coronavirus (the SARS-CoV-2 virus) emerged, which spread fast across the world, and has led to a pandemic. The disease caused by this virus, called COVID-19, has a mild course in a high number of infected people, but is known to have a more severe course in some. Currently, there are no successful treatments with a known effect on the course of the disease in patients suffering from COVID-19. In this study, we will examine whether plasma, a treatment that has been used in human subjects for other diseases (and is known to be safe), can be used to influence the course of COVID-19 towards a lower severity.

The aim of the study is to evaluate clinical efficacy and safety of convalescent plasma for COVID-19.

This clinical trial is an adaptive, randomized, open-label phase II proof-of-concept study to investigate the safety and effect of potentially interesting treatments, for the treatment of hospitalized adult patients suffering from COVID-19.

Because an active treatment for COVID-19 is lacking, plasma donation is now being proposed. To investigate this effect of plasma, we will compare two groups of patients. One group will get standard treatment, plus plasma from a patient recently cured from COVID-19. A second group will get standard treatment alone. In this study, 2 patients out of 3 will receive plasma, and 1 patient out of 3 will receive standard treatment alone. After the study, we will be able to establish whether plasma donation is useful or not.

ELIGIBILITY:
Inclusion Criteria:

1. Subject (≥18 years old) or legally authorized representative provides informed consent prior to initiation of any study procedures.
2. Subject (or legally authorized representative) understands and agrees to comply with planned study procedures.
3. Male or non-pregnant female adult ≥18 years of age at time of enrolment.
4. Patient should be hospitalized
5. Has a confirmed diagnosis of SARS-CoV-2 infection, defined as either:

   1. laboratory-confirmed SARS-CoV-2 infection as determined by PCR, or other commercial or public health assay in any specimen as diagnosed within 60 hours prior to randomization or
   2. The combination of upper or lower respiratory infection symptoms (fever, cough, dyspnea, desaturation) and typical findings on chest CT scan and absence of other plausible diagnoses
6. Illness of any duration, and at least one of the following:

   1. Radiographic infiltrates by imaging (chest x-ray, CT scan, etc.), or
   2. Clinical assessment (evidence of rales/crackles on exam) AND SpO2 ≤ 94% on room air, or
   3. Requiring supplemental oxygen.
7. ABO D typing of the patient should be done at least once and the result should be known.

Exclusion Criteria:

1. Receiving invasive (any mode where a patient has been intubated endotracheally, or via tracheostomy) or non-invasive (for instance, but not restricted to CPAP, PSV, PCV, SiMV) mechanical ventilation before or upon randomization.
2. Pregnancy or breast feeding.
3. Any medical condition which would impose an unacceptable safety hazard by participation to the study.
4. Patients with a documented grade 3 allergic reaction after the administration of fresh frozen plasma (i.e. systemic reaction with cardiovascular and/or respiratory involvement)
5. Patients that have treatment restriction that excludes mechanical ventilation and/or endotracheal intubation
6. Rituximab or another anti-CD20 monoclonal antibody (f.ex. obinutuzumab) has been administered during the year prior of the date of admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 483 (Actual)
Dates: Start 2020-05-02 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Patients requiring mechanical ventilation or death | No mechanical ventilation at day 15 after hospitalization.
  Primary outcome of the study is the number of patients alive without mechanical ventilation at day 15 after hospitalization.

SECONDARY OUTCOMES:
Clinical status of subject at day 15 and day 30 (on a 10-point "WHO progression" ordinal scale) | day 15 and day 30
  0. Uninfected. Non viral RNA detected
  1. Ambulatory, Asymptomatic, viral RNA detected
  2. Ambulatory, Symptomatic, Independent
  3. Ambulatory, Symptomatic, Assistance needed
  4. Hospitalized, mild disease, No oxygen therapy needed
  5. Hospitalized, mild disease, Oxygen by mask of nasal prongs
  6. Hospitalized, severe disease, Oxygen by NIV or High flow
  7. Hospitalized, severe disease, Intubation and mechanical ventilation (pO2/FiO2>=150 OR SpO2/FIO2>=200)
  8. Hospitalized, severe disease, Mechanical ventilation (pO2/FiO2<150 OR SpO2/FIO2<200) OR vasopressors (norepinephrine >0.3 microg/kg/min)
  9. Hospitalized, severe disease, Mechanical ventilation pO2/FiO2<150 AND vasopressors (norepinephrine >0.3 microg/kg/min), OR Dialysis OR ECMO
  10. Death, Dead

CONTACTS AND LOCATIONS:
Overall Officials: Geert Meyfroidt, MD, PhD, Study Director — UZ Leuven
Locations (21):
- Belgium (21):
  - ZNA, Antwerp
  - Imelda Ziekenhuis Bonheiden, Bonheiden
  - Institut Bordet, Brussels
  - UMC Sint-Pieter, Brussels
  - CHU Brugmann, Brussels
  - Erasmus Ziekenhuis, Brussels
  - UZ Brussel, Brussels
  - Cliniques Universitaires St Luc, Brussels
  - AZ Sint-Vincentius, Deinze
  - AZ Maria Middelares, Ghent
  - AZ Sint-Lucas, Ghent
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - CHC Liège Mont Légia, Liège
  - CHR Citadelle Liège, Liège
  - CHU Liège Sart-Tilman, Liège
  - CHU Ambroise Paré, Mons
  - CHR Jolimont Mons-Hainaut, Mons
  - AZ Delta, Roeselare
  - Sint-Trudo Ziekenhuis, Sint-Truiden
  - Centre Hospitalier de Wallonie Picarde (CHwapi), Tournai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Devos T, Geukens T, Schauwvlieghe A, Arien KK, Barbezange C, Cleeren M, Compernolle V, Dauby N, Desmecht D, Grimaldi D, Lambrecht BN, Luyten A, Maes P, Moutschen M, Romano M, Seyler L, Nevessignsky MT, Vandenberghe K, van Griensven J, Verbeke G, Vlieghe E, Yombi JC, Liesenborghs L, Verhamme P, Meyfroidt G. A randomized, multicentre, open-label phase II proof-of-concept trial investigating the clinical efficacy and safety of the addition of convalescent plasma to the standard of care in patients hospitalized with COVID-19: the Donated Antibodies Working against nCoV (DAWn-Plasma) trial. Trials. 2020 Nov 27;21(1):981. doi: 10.1186/s13063-020-04876-0. PMID 33246499

DOCUMENTS (2):
  • Study Protocol (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/54/NCT04429854/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT04429854/SAP_001.pdf